CLINICAL TRIAL: NCT07342127
Title: Evaluation of a Preventive Therapeutic Strategy for Postpartum Venous Thromboembolism in Asymptomatic Women With Heterozygous Factor V Leiden ou Factor II Mutation.
Brief Title: Evaluation of a Preventive Therapeutic Strategy for Postpartum Venous Thromboembolism in Women With Genetic Risk Factor
Acronym: POSTPART AS5-2
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL25_1157; 2025-A02800-49 (Other: ID-RCB)
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Factor V Leiden Heterozygous Mutation; Factor II Heterozygous Mutation; Pregnancy; Postpartum
Keywords: Veinous thromboembolism (VTE); Pregnancy; Postpartum; Thromboprophylaxis; Heterozygous factor V Leiden mutation; Prothrombin gene mutation; Thrombophilia; Low molecular weight heparin (LMWH)
MeSH Terms: conditions — Thrombophilia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 2 weeks or less postpartum thromboprophylaxis: Patients receiving 2 weeks (or less) preventive anticoagulation with low molecular weight heparin after giving birth
  Interventions: Other: Retrospective collection of health data; Other: Phone call to every participant
- 6 weeks postpartum thromboprophylaxis: Patients receiving 6 weeks preventive anticoagulation with low molecular weight heparin after giving birth
  Interventions: Other: Retrospective collection of health data; Other: Phone call to every participant

INTERVENTIONS:
Other: Retrospective collection of health data — From Hospices Civils de Lyon database, collection in Word Excel document of anonymized health data :
  Age, contact details, medical history, first degree family medical history, smoking status, previous estroprogestative contraception utilization, number of gestation, number of miscarriages, any medically assisted reproduction, singleton ou multiple pregnancy, obstetrical complication such as preeclampsia or postpartum hemorrhage, due date, delivering mode, any procoagulant treatment administration, anesthesia, thromboprophylaxis treatment duration
Other: Phone call to every participant — Phone call to every participant to assess any thromboembolic event in 12 first postpartum weeks, any treatment side effect, and their personal experience of the treatment

SUMMARY:
Background : pregnancy and postpartum period are times of increased risk for deep vein thrombosis (DVT).

The incidence of venous thromboembolic disease (VTE) during pregnancy is estimated at 1-2 per 1,000, and this risk increases in the postpartum period, rising up to 80-fold. VTE is a multifactorial condition, and several studies have identified risk factors for DVT during this period. These factors may be related to the patient herself-such as age, overweight, smoking, a personal or family history of DVT, and/or thrombophilia. Factors related to the pregnancy itself and peripartum events-such as preeclampsia, multiple pregnancy, the mode of delivery (emergency or elective cesarean section), and postpartum hemorrhage-have also been identified as DVT risk factors.

Resistance to activated protein C caused by the Factor V Leiden mutation affects about 5% of the population and, in its heterozygous form, increases the risk of VTE by 3- to 10-fold depending on the study, raising the absolute risk to approximately 1 in 400. The heterozygous mutation of the prothrombin (Factor II) gene affects about 2% of the population and increases the risk of VTE threefold. However, although the risk is increased, the absolute risk of VTE remains low (0.5 to 1%).

Regarding prevention, recommendations are heterogeneous and often based on a low level of evidence. In certain situations (e.g., history of provoked thrombosis, moderate thrombophilia), prophylaxis is not always recommended, or its duration is not clearly defined, and the benefit-risk balance remains uncertain.

The main objective of this study is to describe the duration of anticoagulation prescribed after delivery according to the characteristics of patients carrying these mutations and their mode of delivery. The secondary composite objective is to compare two treatment durations (less than 2 weeks vs. 6 weeks) to determine whether a shorter treatment is less effective in preventing deep vein thrombosis, and whether a longer treatment is associated with more adverse effects.

The target population therefore consisted of adult women carrying an asymptomatic heterozygous mutation of Factor V or Factor II, who had been followed up or had consulted at the Hospices Civils de Lyon for obstetric or hematologic evaluation related to this mutation.

Investigators extracted health data of the included patients from the Hospices Civils de Lyon medical software. They also contacted patients by phone to complete data collection, particularly to determine whether they had experienced a deep vein thrombosis within 12 weeks after delivery, or any adverse effects related to anticoagulant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Heterozygous asymptomatic Factor V Leiden mutation or Factor II mutation, diagnosed before or during pregnancy
* Delivering between 01/01/2020 and 31/12/2025
* Patient with French social security rights

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients over than 18 years old, carrying asymptomatic heterozygous Factor V Leiden or Factor II mutation ; who consulted in Hospices Civils de Lyon for this condition, and who delivered between 01/01/2020 and 31/12/2026.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Thromboprophylaxis treatment duration | At baseline
  Evaluation of the given thromboprophylaxis treatment duration according to patients' characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Rugeri, Principal Investigator — Service de Gynécologie Obstétrique - Hôpital de la Croix Rousse
Locations (2):
- France (2):
  - Service d'hémostase clinique - Hôpital Louis Pradel, Bron
  - Service Gynécologie Obstétrique - Hôpital de la Croix Rousse, Lyon